CLINICAL TRIAL: NCT03030469
Title: A Cluster-randomized Trial of Modifying Electronic Health Record Defaults to Reduce the Prescribed Quantity of Opioid Analgesics in Dentistry Practices
Brief Title: Electronic Defaults to Reduce Opioid Prescribing in Dentistry Practices
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: Albert Einstein College of Medicine (Other)
Responsible Party: Principal Investigator, Marcus Bachhuber, Assistant Professor, Montefiore Medical Center
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2016-7373
Record Dates: First submitted 2016-12-19; First posted 2017-01-25 (Estimated); Last update posted 2018-08-14 (Actual); Status verified 2018-08

CONDITIONS: Acute Pain
MeSH Terms: conditions — Acute Pain

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (3):
- 10-pill default (Experimental): The intervention condition consists of a change to the electronic health record so that new opioid analgesic prescriptions automatically default to 10 pills (i.e., the "quantity dispensed" field is pre-populated). This value is modifiable by providers who can tailor the prescription based on clinical factors.
  Interventions: Other: Change in electronic health record default for new opioid analgesic prescriptions
- 5-pill default (Experimental): New opioid analgesic prescriptions will automatically default to 5 pills.
  Interventions: Other: Change in electronic health record default for new opioid analgesic prescriptions
- Standard of care (No Intervention): The control condition will be the usual electronic health record interface. The default number of pills varies by medication, most medications currently have either a blank default or a default of 30 pills.

INTERVENTIONS:
Other: Change in electronic health record default for new opioid analgesic prescriptions
  Arms: 10-pill default; 5-pill default

SUMMARY:
The goal of this research is to investigate the impact of changing opioid analgesic prescribing defaults on the quantity of opioids prescribed for acute non-cancer pain in adult dentistry settings. We will change prescribing defaults for select short-acting opioid analgesics including immediate release oxycodone and hydrocodone as well as codeine and tramadol, including their co-formulations with acetaminophen. In a cluster-randomized trial of three Montefiore Medical Center dentistry sites, we will evaluate the impact of this intervention on patient-level outcomes using 18 months of data (6 months pre-intervention and 12 months post-intervention).

ELIGIBILITY:
Clinical Site Inclusion Criteria:

* Dentistry clinic within Montefiore Medical Center

Patient Inclusion Criteria:

* Received a new opioid analgesic prescription, defined as no opioid analgesic prescription in the preceding 6 months

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10000 (Estimated)
Dates: Start 2016-12; Primary Completion 2018-07-13 (Actual); Study Completion 2018-07-13 (Actual)

PRIMARY OUTCOMES:
Initial prescription number of pills to dispense | Through study completion (18 months)
  From the electronic health record

SECONDARY OUTCOMES:
Initial prescription morphine milligram equivalents to dispense | Through study completion (18 months)
  From the electronic health record
Opioid analgesic reorder (y/n) | Within 30 days after the initial prescription
  From the electronic health record
Total opioid analgesic pills to dispense, including re-orders | Within 30 days after the initial prescription
  From the electronic health record
Total morphine milligram equivalents to dispense, including re-orders | Within 30 days after the initial prescription
  From the electronic health record
Outpatient visits | Within 30 days after the index prescription
  From the electronic health record
Emergency department visits | Within 30 days after the initial prescription
  From the electronic health record
Hospitalizations | Within 30 days after the initial prescription
  From the electronic health record

CONTACTS AND LOCATIONS:
Overall Officials: Marcus Bachhuber, MD, Principal Investigator — Montefiore Medical Center

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bachhuber MA, Nash D, Southern WN, Heo M, Berger M, Schepis M, Sugarman OK, Cunningham CO. Reducing Opioid Analgesic Prescribing in Dentistry Through Prescribing Defaults: A Cluster-Randomized Controlled Trial. Pain Med. 2023 Jan 4;24(1):1-10. doi: 10.1093/pm/pnac106. PMID 35792881